CLINICAL TRIAL: NCT01723722
Title: Treatment of Neonatal Abstinence Syndrome: Evaluation of Efficacy of Phenobarbital in Combination With Either Methadone or Diluted Deodorized Tincture of Opium as Stabilizing and Tapering Regiments
Brief Title: Treatment of Neonatal Abstinence Syndrome
Acronym: HOMENOW
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eastern Maine Medical Center (Other)
Responsible Party: Principal Investigator, Mark S Brown, MD, Chief of Pediatric Service, Neonatalogy, Eastern Maine Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-2-M-107
Record Dates: First submitted 2011-01-27; First posted 2012-11-08 (Estimated); Results first posted 2013-11-27 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Neonatal Abstinence Syndrome
Keywords: Neonatal Abstinence Syndrome; Methadone; Diluted Deodorized Tincture of Opium; dDTO; Phenobarbital
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Phenobarbital and Methadone) (Active Comparator): The following is a dosing guide for methadone:
  1. The neonatal concentration is 1 mg/ml of methadone. It is administered orally every 12 hours.
  2. For the first 24 hours, doses will be prescribed every 6 hours using a sliding scale in response to the last NAS score:
     NAS Score Methadone dose 8-11 0.05 mg/kg/dose 12-15 0.1 mg/kg/dose
     ≥16 0.15 mg/kg/dose
  3. Maximum dose of methadone will be 0.15 mg/kg/dose.
  4. After the first 24 hours of treatment, the total methadone dose will be summed and that dose divided into two doses, given 12 hours apart. For the following 24 hours, additional doses may be given every 6 hours as needed and added to the next 24 hour's doses divided every 12 hours, until NAS scores are consistently <8 for 48 hours.
  5. If at any pointthe maximum dose of methadone is reached and withdrawal is not controlled, then in the opinion of two neonatologists the patient can be crossed-over to the dDTO arm.
  Interventions: Drug: Methadone
- 2 (Phenobarbital and Diluted Deodorized Tincture of Opium) (Active Comparator): The following is a dosing guide for dDTO:
  1. The neonatal concentration is 1:24 dilution for a concentration of 0.4%, equivalent to 0.4 mg/ml of morphine. It is administered orally every 4 hours.
  2. The starting dose will be determined using a sliding scale in response to the last NAS score before starting.
     NAS Score Starting dDTO dose 8-11 0.4 mg/kg/day 12-15 0.6 mg/kg/day
     ≥16 0.8 mg/kg/day
  3. The maximum dose of DTO will be 0.8 mg/kg/day.
  4. After the first 24 hours of treatment, if the NAS scores are still ≥8, the dose will be increased to the next level.
  5. If at any point the maximum dose of methadone is reached and withdrawal is not controlled, then in the opinion of two neonatologists the patient can be crossed-over to the methadone arm.
  Interventions: Drug: Diluted Deodorized Tincture of Opium

INTERVENTIONS:
Drug: Methadone — Concentration is 1mg/mL administered every 12 hours given on sliding scale in response to last NAS score.
  Other Names: Dolophine
  Arms: 1 (Phenobarbital and Methadone)
Drug: Diluted Deodorized Tincture of Opium — Concentration is 1:24 dilution for a concentration of 0.4%
  Other Names: Laudanum
  Arms: 2 (Phenobarbital and Diluted Deodorized Tincture of Opium)

SUMMARY:
This study compares treatment of Neonatal Abstinence Syndrome (NAS) with two different drugs for the difference in the length of treatment. This is a randomized, open-label comparison of phenobarbital and methadone versus phenobarbital and diluted deodorized tincture of opium (dDTO) where phenobarbital is the initial drug used to stabilize neonatal withdrawal.

DETAILED DESCRIPTION:
a.Procedures: NAS scoring is currently done on infants meeting the inclusion criteria [IDD 29:070]. NAS scores are initially done every 2 hours for 24 hours and then every 4 hours when awake or before feeding for the duration of observation or treatment.

i. NAS scores may indicate more than withdrawal. Conditions such as colic, reflux, or baseline irritability may influence the baseline scores. Decisions made based on the NAS scores should take into account these factors and the baseline for the infant.

b.Emergence of symptom, dosing, and initiation of treatment: Withdrawal is defined as at least 2 NAS scores >8 or 1 NAS score >12. Once withdrawal has emerged, the infant will be given: i. Phenobarbital 20 to 30 mg/kg to load divided in up to 3 doses over 24 hours and maintenance phenobarbital should be started at 2.5 mg/kg/dose administered Q 12h, 12 hours after the loading dose is ended. NAS scoring is continued and if scores remain <8 for a minimum of 5 days after starting phenobarbital, the infant is eligible for discharge.

ii. If after phenobarbital treatment has been started, at least 2 NAS scores >8 or 1 NAS score >12, then a phenobarbital level will be drawn and a mini-load calculated to reach a level of 30 mg/dl. If withdrawal is not controlled or re-emerges after the mini-load dose, the infant will be randomized to one of the two arms of the study - methadone or dDTO.

iii. Twins will be randomized together to the same arm. iv. Randomization will be stratified into mothers on narcotic treatment >3 months and those not in treatment or <3 months. Randomization will be done in blocks of 10 for each stratum.

v. For both drugs, the neonatal preparation will be used. vi. The following is a dosing guide for methadone:

1. The neonatal concentration is 1 mg/ml of methadone. It is administered orally every 12 hours - standardized eventually to 0900 and 2100.
2. For the first 24 hours, doses will be prescribed every 6 hours for 4 doses, using a sliding scale in response to the last NAS score:

   NAS Score Methadone dose 8-11 0.05 mg/kg/dose 12-15 0.1 mg/kg/dose >16 0.15 mg/kg/dose
3. Maximum loading dose of methadone will be 0.15 mg/kg/dose Q 6 hour
4. After the first 24 hours of treatment, the total methadone dose will be summed and that dose divided into two doses, given 12 hours apart. Subsequently, PRN doses of 0.05 mg/kg/dose may be given every 6 hours for scores >8 X 2 and added to the next 24 hour's doses, divided every 12 hours, until NAS scores are consistently <8 for 48 hours.
5. If at any point the maximum dose of methadone is reached and withdrawal is not controlled, then in the opinion of two neonatologists the patient can be crossed-over to the dDTO arm.

vii. The following is a dosing guide for dDTO:

1. The neonatal concentration is 1:24 dilution for a concentration of 0.4%, equivalent to 0.4 mg/ml of morphine. It is administered orally every 4 hours - standardized eventually to 0400, 0800, 1200, 1600, 2000, 0000.
2. The starting dose is determined by using a sliding scale in response to the last NAS score before starting:

   NAS Score dDTO dose 8-11 0.1 mg/kg/day 12-15 0.15 mg/kg/day >16 0.2 mg/kg/day

   For next day, the maintenance dose will return to the previous dose and given in 6 divided doses given Q 4 hours.

   iv. For either methadone or dDTO, dosing will be held at this level and weaning will be resumed when the infant has NAS scores <8 for 48 hours.

   e. Holding of doses: Methadone or dDTO will be held for poor feeding, respiratory depression, or somnolence at any time in the protocol.

   f. Behavioral assessment: Behavioral assessment will be done by two methods. The first by actigraphy and the second by NINS, both during the second week of weaning. The latter will be done prior to a scheduled phenobarbital dose.

   g. Formula: A 24 kcal/ounce formula should be fed initially using either standard formula or by adding breast milk fortifier. During the weaning period, when weight gain is >30 grams/day for at least 2 days, formula will be changed to 20 kcal/ounce and weight gain monitored. If not sustained, then formula should be changed back to 24 kcal/ounce.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of opioid withdrawal clinically as defined by 2 NAS scores >8 or 1 NAS score >12 over a 4 to 8 hour time period, AND
* Gestation >=35 weeks at entry defined by best obstetrical and physical exam criteria, AND
* Medically stable condition, other than in opioid withdrawal, in the opinion of the attending neonatologist, AND EITHER,
* Meconium or urine drug screen positive for opioids on mother or newborn, OR
* Known maternal prescription of opioids for chronic pain management during at least the last trimester of pregnancy, OR
* Known maternal prescription of opioids for treatment of addiction, OR
* Suspected or admitted abuse with opioid drugs
* Infants of mothers with a medical or psychiatric diagnosis will not be excluded, unless the maternal diagnosis precludes informed consent

Exclusion Criteria:

* Gestation <35 weeks at entry defined by best obstetrical and physical exam criteria.
* Hypoglycemia, hypomagnesaemia, or hypocalcaemia until corrected.
* Serious medical illness such as sepsis, pneumonia, hyperthyroidism, meningitis, intracranial hemorrhage, perinatal depression, or respiratory failure requiring admission to the NICU.
* Evidence of major congenital anomalies or genetic syndromes that impact the neonatal course.

Ages: 1 Day to 6 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2007-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark S. Brown, MD, Principal Investigator — Eastern Maine Medical Center
Locations (1):
- Eastern Maine Medical Center, Bangor, Maine, United States

REFERENCES:
- [Derived] Zankl A, Martin J, Davey JG, Osborn DA. Opioid treatment for opioid withdrawal in newborn infants. Cochrane Database Syst Rev. 2021 Jul 7;7(7):CD002059. doi: 10.1002/14651858.CD002059.pub4. PMID 34231914

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period 11/15/2007 through 9/1/2009; location Eastern Maine Medical Center NICU
Pre-assignment Details: Exclusion for other medical conditions causing withdrawal symptoms, gestation less than 35 weeks
Groups:
- Methadone After Phenobarbital for Withdrawal: for withdrawal reaching treatment threshold phenobarbital was first started and if a second drug was needed randomization was done after consent; this arm started methadone
- Deodorized Tincture Opium After Phenobarbital for Withdrawal: for withdrawal reaching treatment threshold phenobarbital was first started and if a second drug was needed randomization was done after consent; this arm started dilute deordorized tincture of opium
Period: Overall Study
Arm/Group | Methadone After Phenobarbital for Withdrawal | Deodorized Tincture Opium After Phenobarbital for Withdrawal
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- DTO After Phenobarbital for Withdrawal: for withdrawal reaching treatment threshold phenobarbital was first started and if a second drug was needed randomization was done after consent; this arm started dilute deordorized tincture of opium
- Total: Total of all reporting groups
Arm/Group | Methadone After Phenobarbital for Withdrawal | DTO After Phenobarbital for Withdrawal | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 20 | 40
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 0.005 (0) | 0.005 (0) | 0.005 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 11 | 12 | 23
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Length of Treatment With Opioid Medication
Description: Up to 12 months
Time Frame: Up to 12 months
Population: Completion of treatment
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Deodorized Tincture Opium After Phenobarbital for Withdrawal | Methadone After Phenobarbital for Withdrawal
Number analyzed (Participants) | 20 | 20
days | 19.1 (8.8) | 17.7 (10)

ADVERSE EVENTS:
Arm/Group | Methadone After Phenobarbital for Withdrawal | DTO After Phenobarbital for Withdrawal
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes